CLINICAL TRIAL: NCT04661436
Title: Multimodal Imaging Evaluation System of Axillary Lymph Node Staging and Treatment Strategy for Breast Cancer Neoadjuvant Therapy
Acronym: MIES-BCNAT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Jun Luo, Principal researchers, Sichuan Provincial People's Hospital
Other Study IDs: MIES-BCNAT
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer; axillary lymph nodes; neoadjuvant therapy; Evagination
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Contrast-Enhanced Ultrasound — The research will study the qualitative analysis indicators of contrast-enhanced ultrasound, including: enhancement uniformity, enhanced range, presence or absence of enhancement defect area, presence or absence of nourishing blood vessels, etc.; and quantitative analysis indicators, including: peak time, peak intensity, rising slope, Area under the curve, etc., analyze the correlation between the changes of various parameters before and after neoadjuvant treatment（NAT） and the pathological response of patients, and try to find indicators and cut-off values that can predict and early evaluate the efficacy.
  This study will study the qualitative and quantitative parameters of MRI-enhanced scanning and the changes of DWI parameters, analyze the correlation between the parameters of patients before and after NAT and pathological response, and try to find indicators and cut-off values that can predict and early evaluate the efficacy.
  Other Names: Magnetic Resonance Imaging

SUMMARY:
In view of the lack of systematic curative effect prediction and early evaluation indicators for breast cancer neoadjuvant chemotherapy, the effective fusion of CEUS（contrast-enhanced ultrasound） and MRI is realized, and a multi-modal standardized evaluation system of NAT based on the dynamics across time and full cycle is constructed, in order to find the predictive effect and early evaluation of NAT. Means to improve the accuracy of NAT patient selection, treatment course selection, and efficacy evaluation, to achieve controllable and individualized and precise NAT, thereby improving efficacy, reducing unnecessary treatment adverse reactions, guiding pathological materials, reducing medical costs, and ultimately improving breast cancer The patient's DFS and OS. In addition, for patients with axillary lymph node cN0 before and after neoadjuvant or descending after neoadjuvant, the evaluation system is used to explore the feasibility, safety, and effectiveness of replacing sentinel lymph node biopsy or carrying out sentinel lymph node biopsy, which is a useful strategy for axillary lymph node management in such patients. Develop a theoretical foundation.

ELIGIBILITY:
Inclusion Criteria:

1. Age and gender: 18 to 70 years old, female;
2. ECOG systemic state 0~1;
3. Screening examinations, including medical history, vital signs measurement, general physical examination, laboratory examinations (blood routine, urine routine, blood biochemistry, blood electrolytes, full set of pre-transfusion, etc.), electrocardiogram, heart and abdomen color Doppler ultrasound, head, chest, Abdominal CT and bone scan to determine whether the subjects are in good health and have distant metastases;
4. According to the RECIST1.1 standard, at least one measurable lesion exists;
5. Invasive breast cancer confirmed by preoperative biopsy pathological examination, clinical stage is II-III [cT2 and any N, cT3 and any N; cT4 and any N, according to the American Joint Committee on Cancer (AJCC) standard] Breast cancer patients;
6. The functional level of organs must meet the following requirements:

   1. Blood routine ANC≥1.5×10 9/L; PLT≥90×10 9/L; Hb≥90 g/L;
   2. Blood biochemistry TBIL≤1.5×ULN; ALT and AST≤2×ULN; BUN and Cr ≤1.5×ULN and creatinine clearance ≥50 mL/min (Cockcroft-Gault formula);
   3. Heart color Doppler ultrasound LVEF≥50%;
   4. 12-lead ECG Fridericia method corrected QT interval (QTcF) female <470 ms.
7. Patients with known hormone receptor status.
8. Patients with negative serum pregnancy tests and patients with reproductive potential must agree to use effective non-hormonal contraceptive methods during treatment and at least 6 months after the last use of the test drug.
9. During the trial period and within 6 months after the trial, female subjects should take medically acceptable or reliable contraceptive measures;
10. Subjects understand the test procedures, voluntarily comply with the requirements of the test protocol, and agree to participate in the test by signing an informed consent form approved by the ethics committee of the participating center.

Exclusion Criteria:

1. Allergic physique, those who are known to be allergic to the components of the test drug (inquiry); those who have a history of allergies to ultrasound contrast agents (sulfur hexafluoride microbubbles) and any contrast agent in enhanced magnetic resonance (inquiry) ；
2. Inflammatory breast cancer; metastatic breast cancer (stage IV)
3. A history of immunodeficiency, including a positive HIV test, or other acquired or congenital immunodeficiency and a history of organ transplantation;
4. Have ever suffered from any heart disease, including: 1) angina pectoris; 2) arrhythmia requiring medication or clinical significance; 3) myocardial infarction; 4) heart failure; 5) any person judged to be unsuitable Other heart diseases participating in this trial.
5. Female patients during pregnancy and lactation, female patients with fertility and a positive baseline pregnancy test, or female patients of childbearing age who are unwilling to take effective contraceptive measures during the entire trial period.
6. According to the judgment of the investigator, there are concomitant diseases that seriously endanger the safety of the patient or affect the completion of the study (including but not limited to severe hypertension that cannot be controlled by drugs, severe diabetes, active infection, etc.).
7. Have a clear history of neurological or mental disorders, including epilepsy or dementia.
8. Any other situation that the researcher considers inappropriate to participate in this research.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Invasive breast cancer confirmed by preoperative biopsy pathological examination, clinical stage is II-III.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantitative analysis parameters and cut-off values of contrast-enhanced ultrasound prediction and early evaluation of NAT efficacy; | Estimated up to 2 year
  By studying the qualitative analysis indicators of contrast-enhanced ultrasound, including: enhancement uniformity, enhanced range, presence or absence of enhancement defect area, presence or absence of nourishing vessels, etc.; and quantitative analysis indicators, including: peak time, peak intensity, rising slope, under the curve Area, etc., analyze the correlation between the changes of the parameters before and after NAT and the pathological response.
Enhanced MRI prediction and DWI for early evaluation of NAT efficacy, and enhanced quantitative analysis parameters and cut-off values | Estimated up to 2 year
  By studying the qualitative and quantitative parameters of MRI-enhanced scanning and the changes of DWI parameters, the correlation between the parameters before and after NAT and the pathological response of patients is analyzed.
Able to predict and assess the stage of axillary lymph nodes after NAT and guide the development of diagnostic criteria for treatment strategies | Estimated up to 2 year
  Combining the high sensitivity of ultrasound in the recognition of superficial lymph nodes, the feasibility of contrast-enhanced ultrasound in the identification, location and diagnosis of sentinel lymph nodes in breast cancer, and the integrity of MRI, to discuss the formulation of multi-imaging systems for the treatment of axillary lymph nodes in patients with lymph node degeneration after NAT The feasibility, safety and effectiveness of clinical application.
Construct a multi-modal and multi-parameter evaluation system and its standards that can predict and early evaluate the efficacy of NAT. | Estimated up to 2 year
  Based on the above three research results, a mathematical model is established, a multi-modal and multi-parameter evaluation system combining multiple images is constructed, and the strengths are complemented to establish an economic and efficient evaluation index system and standardized process.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Luo, Master, Principal Investigator — Sichuan Provincial People's Hospital; Jie Chen, Master, Study Director — Sichuan Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: No